CLINICAL TRIAL: NCT05376007
Title: The Effectiveness of the Serious Game 'Broodles' in Improving Psychosocial Well-being of Siblings (6-9 Years Old) of Children With Visual Impairment and/or Intellectual Disability: A Randomized Controlled Trial
Brief Title: Effectiveness of the Serious Game 'Broodles' for Siblings of Children With Visual Impairment and/or Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, prof. dr. Paula S. Sterkenburg, Endowed professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL79852.029.22; NL79852.029.22 (Registry Identifier: CCMO)
Record Dates: First submitted 2022-04-21; First posted 2022-05-17 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: siblings; visual impairment; intellectual disability; quality of life; well-being
MeSH Terms: conditions — Vision Disorders; Intellectual Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and investigators will be masked at pre-test assessment only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Playing serious game 'Broodles' (Experimental): The participants allocated to this group will play the newly developed serious game 'Broodles' after pre-test assessment. Children will play the serious game without the parent or the help of a caregiver. Parents and children will make complementary worksheets together and parents will read an information brochure.
  Concomitant care as usual is allowed during the study.
  A parent-child pair is labelled as one participant.
  Interventions: Behavioral: Serious game 'Broodles'
- Waitlist control group (No Intervention): The participants allocated to this group will play the serious game 'Broodles' after follow-up assessment.
  Concomitant care as usual is allowed during the study.

INTERVENTIONS:
Behavioral: Serious game 'Broodles' — The serious game 'Broodles' is a newly developed web-based, educational game that can be played by siblings on a computer or tablet without support from an adult. The game discusses the nine domains of sibling quality of life (Moyson & Roeyers, 2012) in eight 20-minute levels. The main characters of the game are the Broodles, which are little monster creatures that experience things that siblings of children with ID and/or VI can also experience. The game includes animations, videos of siblings talking about their experiences, quizzes and mini-games. These elements are focussed on emotions, thoughts and difficult situations that siblings can experience. In addition to the game, siblings make offline worksheets and parents receive an information brochure. Siblings complete the game in four weeks.
  Arms: Playing serious game 'Broodles'

SUMMARY:
The support for siblings of children with disabilities is scarce and fragmented, even though studies have shown that these siblings can benefit from support. Although some interventions for siblings have been developed, these are costly and time-consuming and the effects have not been researched thoroughly with randomized controlled trials. This study will investigate the effectiveness of the newly developed serious game 'Broodles' in improving the quality of life and psychosocial well-being of healthy siblings (aged 6-9 years) of children with intellectual disability (ID) and/or visual impairment (VI). The effectiveness of the serious game will be examined in a randomized controlled trial (RCT) with a pre-test (T0), post-test (T1) and follow-up (T2). There will be two groups, namely an experimental group playing the serious game and a waitlist control group. Quantitative and qualitative measures will be used including questionnaires, drawings and open-ended questions. Both the sibling and one parent will complete the assessments.

The serious game, named 'Broodles', is a psychological intervention that addresses how to handle thoughts and emotions concerning several important issues in the lives of siblings. The game has 8 levels that take approximately 20 minutes to play. In addition to the serious game, children make offline worksheets and parents receive tips and information on how to support their child. The primary study parameters are quality of life and sibling adjustment to and perceptions of the disability of the brother or sister. Secondary study parameters are different aspects of psychosocial well-being, including self-esteem, experienced social support, sibling relationship, coping skills, parent-child relationship, and social validity. It is expected that the participants in the experimental conditions will benefit from playing the game, namely their quality of life and psychosocial well-being is expected to improve.

DETAILED DESCRIPTION:
A detailed description can be found in the published protocol in Trials.

ELIGIBILITY:
Inclusion Criteria:

* Having a brother or sister with (strongly suspected) visual impairment and/or intellectual disability (0-17;11years old), with possibly other comorbid disabilities, disorders or illnesses.
* The brother or sister with a disability lives in the same house (at least part of the time)
* Living in the Netherlands or Flanders (Dutch speaking part of Belgium)

Exclusion Criteria:

* Having a disability, impairment or severe illness
* Brother or sister with VI and/or ID lives in a residential care facility on a full-time basis
* One or both parents have a disability, impairment or severe illness
* Not speaking the Dutch language
* No written consent from the participant and/or their legal representative
* Another sibling in the household is already included in the study. Only one sibling per household can participate in the study. The parents will decide which sibling will participate.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Change in quality of life as assessed by the Psychosocial Health Summary Score of the Pediatric Quality of Life Inventory (PedsQL 4.0) - Acute Version - | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  The quality of life of the participating sibling is measured with both a child-report and parent-report version of the questionnaire Pediatric Quality of Life Inventory (PedsQL 4.0) - Acute Version - Psychosocial Health Summary Score. The total score on this scale has a minimum of 0 and a maximum of 60, with a higher score indicating more problems, and thus lower quality of life. The change in score over time on this outcome is measured, with a decreased score indicating improved quality of life.
Change in Sibling adjustment to and perceptions of their brother or sister's disability | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  Sibling adjustment to and perceptions of their brother or sister's disability is measured with both a child-report and parent-report version of the Sibling Perception Questionnaire (SPQ) - Negative Adjustment Scale. The total score on this scale has a minimum of 18 and a maximum of 72, with a higher score indicating more negative adjustment to the disability of the brother or sister. The change in score over time on this outcome is measured, with a decreased score indicating improved adjustment.

SECONDARY OUTCOMES:
Change in Self-esteem | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  The self-esteem of the sibling is measured with the child-report questionnaire Self-Perception Profile for Children simplified(SPPC-s) - Global Self-Worth subscale. The total score on this scale has a minimum of 3 and a maximum of 12, with a higher score indicating higher self-esteem. The change in score over time on this outcome is measured, with an increased score indicating improved self-esteem.
Change in Perceived social support | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  The perceived social support of the participating sibling is measured with the child-report questionnaire Social Support Scale for Children (SSSC). The total score on this scale has a minimum of 24 and a maximum of 96, with a higher score indicating higher perceived social support. The change in score over time on this outcome is measured, with an increased score indicating improved perceived social support.
Change in sibling relationship (child-report) | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  Sibling relationship between the participating sibling and the sibling that has a disability is measured with the child-report drawing task Pictorial Assessment of Interpersonal Relationships (PAIR). This instrument has six separate scales.
  The scales Cohesion and Distancing have total score ranges from 0 to 6, with a higher score indicating respectively higher interdependence and higher autonomy in the relationship.
  The scales Similarity and Value have total score ranges from 0 to 10, with a higher score indicating respectively higher affinity and higher disparity between the siblings.
  The scales Emotion and Conflict have nominal and ordinal scores (1-4), with a higher score indicating respectively more similarity in emotional state and a amore disrupted relationship.
  The change in score over time on this outcome is measured. In addition thematic analysis is executed, and changes in themes over time are measured.
Change in sibling relationship (parent-report) | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  Sibling relationship between the participating sibling and the sibling that has a disability is measured with the parent-report questionnaire Parental Expectations and Perceptions of Children's Sibling Relationships Questionnaire (PEP-SRQ). This scale has three separate subscales.
  These include the scales Warmth (total score ranges from 15 to 80), Agonism (total score ranges from 9 to 45), and Rivalry/Competition (total score ranges from 3 to 15). A higher score indicates respectively more warmth, more agonism, and more rivalry in the sibling relationship as perceived by the parent.
  The scale also has a question about the total quality of the sibling relationship, as perceived by the parent (range 1-7), with a higher score indicating higher quality of the relationship.
  The change in score over time on this outcome is measured.
Change in coping skills | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  Copings skills of the participating sibling are measured with a 12-item version of the child-report questionnaire Coping Strategies Inventory (CSI).Two separate subscales are used: Engaged and Disengaged Coping. The total score on both scales have a minimum of 5 and a maximum of 30. A higher scored on the Engaged scale means higher use of engaged coping strategies. A higher score on the Disenganged scale means higher use of disengaged coping strategies. The baseline change in scores over time on this outcome is measured.
Change in parent-child relationship | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  The parent-child relationship between the participating sibling and the participating parent is measured with the parent-report questionnaire Child-Parent Relationship Scale (CPRS) - Closeness scale, short version.
  The total score on this scale has a minimum of 7 and a maximum of 35, with a higher score indicating a closer parent-child relationship. The change in score over time on this outcome is measured.
Social validity of the intervention | post-test (T1, week 6; only group 1)
  The social validity of the intervention is measured with an adapted version of the child-report and parent-report questionnaire Social Validity Scale (SVS). The mean score on the scale, ranging from 1 to 5, will be used.
Subjective evaluation of the intervention | post-test (T1, week 6; only group 1)
  Participants (both parents and children) answer open-ended evaluation questions about the intervention at post-test assessment. This includes questions about what they think was good about the intervention, what they think could be better, and what they think they learned from the intervention.
Change in Sibling adjustment to their brother or sister's disability | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  Sibling adjustment to their brother or sister's disability is measured with self-developed open ended questions that are answered by the parent and the child. The questions include: (1) "Can you name up to five examples of what you/your child like(s)about your/their brother or sister?" (2) "Can you name up to five examples of what you/your child do(es)not like or find(s)difficult or unpleasant about having a brother or sister with a disability?" (3) "Can you explain what you/your child do(es)to deal with these examples?" The children are also asked to rate the examples named at question 1 and question 2 with smileys (5-point scale), indicating how much they like it or how hard they think it is.
  Thematic analysis is executed, and changes in themes over time are measured. Change over time in smileys is measured as well.

OTHER OUTCOMES:
Change in Parenting self-efficacy as assessed by a 3-item version of the Parenting Sense of Competence Scale (PSOC) | pre-test (T0, week 1), post-test (T1, week 6), follow-up (T2, week 12-14)
  The parenting self-efficacy of the participating parent is measured using a 3-item version of the parent-report questionnaire Parenting Sense of Competence Scale (PSOC). The total score on this scale has a minimum of 3 and a maximum of 15, with a higher score indicating higher parenting self-efficacy. The change in score over time on this outcome is measured, with an increased score indicating improved parenting self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Paula S Sterkenburg, prof. dr., Principal Investigator — VU University of Amsterdam
Locations (1):
- VU University Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized quantitative IPD of the participants that gave additional consent, will be shared with other researchers upon reasonable request. This includes the scores on the following questionnaires: PedsQL, SPQ, SPPC, SSSC, CSI, CPRS and PSOC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The study protocol, including the statistical analysis plan, will be published in Trials (date unknown). The informed consent form, full study protocol and analytic code can be shared upon reasonable request.
Access Criteria: To be determined

REFERENCES:
- [Derived] Veerman LKM, Willemen AM, Derks SDM, Brouwer-van Dijken AAJ, Sterkenburg PS. The effectiveness of the serious game "Broodles" for siblings of children with intellectual disabilities and/or visual impairment: study protocol for a randomized controlled trial. Trials. 2023 May 17;24(1):336. doi: 10.1186/s13063-023-07358-1. PMID 37198687